CLINICAL TRIAL: NCT04914403
Title: A Phase I, Open Label, Dose Escalation Study to Evaluate the Safety and Tolerability After Intravenous Infusion of UMC119-06-05 in Elderly Subjects With Mild to Moderate Frailty Syndrome.
Brief Title: Mesenchymal Stem Cells for The Treatment of Frailty Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMC119-06-05-FS-01
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Frailty Syndrome
Keywords: frailty syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Cohort 1: Low dose of UMC119-06-05 Cohort 1: High dose of UMC119-06-05
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UMC119-06-05 (Experimental): Human Umbilical Cord Derived-Mesenchymal Stem Cells, Single treatment by intravenous infusion.
  Interventions: Biological: UMC119-06-05

INTERVENTIONS:
Biological: UMC119-06-05 — Cohort 1: Low does of UMC119-06-05 Cohort 2: High does of UMC119-06-05

SUMMARY:
The clinical study with UMC119-06-05 is designed to investigate the safety in patients with frailty syndrome. This will be a dose escalation, open label, single-center study in adult with frailty syndrome. UMC119-06-05 is ex vivo cultured human umbilical cord tissue-derived mesenchymal stem cells product which is intended for treatment of frailty syndrome.

DETAILED DESCRIPTION:
Frailty syndrome is the most problematic expression of population ageing and profound implications for the planning and delivery of health and social care when population ageing is accelerating rapidly worldwide, from 461 million people older than 65 years in 2004 to an estimated 2 billion people by 2050 . Frailty syndrome characterized by a progressive decline in health and clinical symptoms of exhaustion, weight loss, a feeling of slowing down, and a decrease in functional capacity. Frailty is a common clinical syndrome in older adults that carries an increased risk for poor health outcomes including falls, incident disability, hospitalization, and mortality. Health study as meeting three out of five phenotypic criteria: low grip strength, self-reported exhaustion, slowed walking speed, low physical activity, and unintentional weight loss. Frailty is a disorder of several inter-related physiological systems, including genetic and environmental factors in combination with epigenetic mechanisms, which regulate the differential expression of genes in cells and could be especially important in ageing. Current interventions focus on interdisciplinary approaches which include nutritional supplementation, physical exercise, and cognitive intervention. Clinical studies of these preventative approaches have shown inconsistent and modest benefits, further highlighting the unmet clinical need. Therefore, development of new therapeutic modalities to improve the clinical outcomes and prognosis of frailty syndrome in adult patients is of urgent need. A variety of pharmacologic and biologic therapies are currently being tested to treat aging. Among the more innovative, experimental therapies, Mesenchymal Stromal Cells (MSCs) are represents an attractive option that addresses the pathophysiology of the syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age between ≥ 60 through ≤ 85 years.
* Subjects show signs of frailty condition as assessed by the Investigator with a Clinical Frailty scale between 4 to 6.
* Subjects with body weight between 40 to 90 kg.
* Subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided.

Exclusion Criteria:

* Subjects unwilling or unable to perform any of the assessments required by endpoint analysis.
* Subjects who have a diagnosis of any disabling neurologic disorder including, but not limited to: Parkinson's disease, Amyotrophic Lateral Sclerosis, multiple sclerosis or dementia.
* Subjects have a score on the Mini-Mental State Examination (MMSE) of 24 or below, or have been unstable on neurological examination within the past 6 months.
* Subjects who have a significant comorbid medical condition(s) including, but not limited to:

  1. Severe kidney disease requiring hemodialysis or peritoneal dialysis;
  2. Advanced liver disease such as hepatitis or liver cirrhosis;
  3. Severe congestive heart failure (NYHA class 3 and 4);
  4. Severe pulmonary dysfunction, including severe chronic obstructive pulmonary disease stage III or IV (Gold classification)
  5. Hypothyroidism (TSH > 10 mU/L) or hyperthyroidism (TSH < 0.1 mU/L)
* Subjects on chronic immunosuppressive transplant therapy.
* Subjects who have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma or in situ carcinomas.
* Subjects using chronic immunosuppressant therapy (including prednisone or equivalent for more than 2 consecutive weeks within the past 3 months) or TNF-alpha antagonists.
* Subjects who are known to be infected with HIV.
* Subjects with known allergy or hypersensitivity to any component of the formulation, including normal saline, human serum albumin, dimethyl sulfoxide (DMSO) and cellular therapies.
* Subjects who have participated in another clinical study of new investigational therapies within 6 months before the study drug administration.
* Subjects have a history of drug or alcohol abuse within the past 3 years.
* Subjects currently in hospital stay.
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.
* Subjects with uncorrected hematology test including, but not limited to:

  1. Hemoglobin < 8 g/dl
  2. White blood cell count < 3,000/mm3
  3. International normalized ratio (INR) of Coagulopathy >1.5
  4. Platelet count < 80,000/mm3
* Subjects who have the following conditions in laboratory tests:

  1. >2 × upper limit of normal for alanine aminotransferase (ALT) or aspartate aminotransferase (AST)
  2. Total bilirubin > 1.5 mg/dl
* Subjects who have a significant illness as judged by principal investigator (PI) including, but not limited to:

  1. Psychiatric illness
  2. Uncontrolled hypertension or hypotension (specify numeric cutoffs)
  3. Unstable cardiac arrhythmia
  4. Severe osteoarthritis or degenerative joint disease
  5. Hepatitis B, Hepatitis C infections
  6. History of COVID-19 in the past 4 weeks or with significant COVID-19 conditions judged by PI, or ongoing COVID-19
* Have any condition that in the opinion of the Principal Investigator limits lifespan to < 1 year.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-06-05. | 3 months from the day of administration
  Incidence of Treatment-Emergent Adverse Events (TEAEs). Incidence of withdrawals due to Adverse Events(AEs).

SECONDARY OUTCOMES:
Changes in exercise performance using 6-min walk test (6MWT). | From baseline up to 360 days after administration.
  The distance (meter) and walking speed (meter per seconds) in a 6-minute walk test. Improvement in clinical function as assessed by mean change in exercise performance using 6-min walk test (6MWT).
Changes in grip strength. | From baseline up to 360 days after administration.
  Hand grip strength can be quantified by measuring the amount of static force that the hand can squeeze around a dynamometer. The force has most commonly been measured in kilograms.
Changes in quality of life measured by change in SF12 (12-Item Short Form). | From baseline up to 360 days after administration.
  The 12-Item Short Form Health Survey (SF-12) is a 12-item measure of perceived health status with good reliability, validity and correlation with other health measures. The score is computed using the scores of the twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Changes in physical activity using International Physical Activity Questionnaire (IPAQ) questionnaire | From baseline up to 360 days after administration.
  The IPAQ calculates the metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. Categorical score to three levels of physical activity are Low, or Moderate, or High.
Changes in Forced Expiratory Volume in One Second (FEV1). | From baseline up to 360 days after administration.
  Improvement in clinical function as assessed by mean change in One Second to the Forced Vital Capacity.
Changes in Clinical Frailty Scale. | From baseline up to 360 days after administration.
  Clinical Frailty Scale evaluates specific domains, including comorbidity, function, and cognition, to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare., New Taipei City, Taiwan